CLINICAL TRIAL: NCT06430658
Title: NEoadjuvant Total RX for Borderline Unresectable Esophageal Squamous Cell Carcinoma: a Prospective Randomized, Three-Arm, Open-Label Phase II Trial (NEXUS-2)
Brief Title: Neoadjuvant Comprehensive Treatment for Unresectable Esophageal Cancer
Acronym: NEXUS-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, YIN LI, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEXUS-2
Record Dates: First submitted 2024-05-13; First posted 2024-05-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Esophagus Cancer
Keywords: Esophagus Cancer; Chemoradiotherapy; conversion surgery; immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ChemoRT+Immuno (Experimental): Surgery was evaluated after chemoradiotherapy (40-41.4Gy/1.8-2Gy/20-23 fractions) followed by two cycles of chemotherapy and immunotherapy.For inoperable patients, immunotherapy was used as maintenance therapy
  Interventions: Combination Product: Tislelizumab (BGB-A317) with chemoradiotherapy
- Immuno+ChemoRT (Experimental): Surgery was evaluated after two cycles of chemotherapy and immunotherapy followed by chemoradiotherapy(40-41.4Gy/1.8-2Gy/20-23 fractions).For inoperable patients, immunotherapy was used as maintenance therapy
  Interventions: Combination Product: Tislelizumab (BGB-A317) with chemoradiotherapy
- ChemoRT (Active Comparator): Surgery was evaluated after concurrent definitive chemoradiotherapy (50-50.4Gy/1.8-2Gy/25-28fractions) .For inoperable patients, immunotherapy was used as maintenance therapy
  Interventions: Combination Product: Tislelizumab (BGB-A317) with chemoradiotherapy

INTERVENTIONS:
Combination Product: Tislelizumab (BGB-A317) with chemoradiotherapy — Different sequences and methods of treatment to convert surgery

SUMMARY:
Patients diagnosed with locally advanced esophageal squamous cell carcinoma (ESCC) that is deemed unresectable face a bleak prognosis. Recent phase 1/2 studies have demonstrated the efficacy and safety of augmenting neoadjuvant concurrent chemoradiotherapy with immunotherapy in treating resectable ESCC. The present study is a prospective, 3-arm, randomized trial that seeks to evaluate the efficacy of diverse conversion therapy modalities in patients with unresectable ESCC. The study objectives include R0 resection rate, treatment-related adverse events, morbidity and mortality, 1-year progression-free survival (PFS), and 1-year overall survival (OS) rates.

Tislelizumab is a humanized IgG4 monoclonal antibody with high affinity/specificity for programmed cell death protein 1 (PD-1). Tislelizumab was specifically engineered to minimize binding to FcɤR on macrophages, thereby abrogating antibody-dependent phagocytosis, a potential mechanism of T-cell clearance and resistance to anti-PD-1 therapy.

This trial will provide valuable insights into the effectiveness of the three conversion therapy modalities and help to inform clinical decision-making for patients with unresectable locally advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed sorely ESCC without other histology subtypes.
2. Thoracic esophageal cancer.
3. No prior anti-cancer treatment, including but not limited to surgery, radiotherapy, chemotherapy, targeted therapy, or immunotherapy.
4. Borderline unresectable locally advanced ESCC deemed by investigators as suspicious of but not confirmed T4b according to the American Joint Committee on Cancer (AJCC) 8th edition staging classification or extracapsular lymph node involvement (ELNI).
5. The Karnofsky Performance Scale (KPS) ≥70.
6. Normal primary organ functions, including but not limited to hemoglobin (Hb) ≥ 100g/L; white blood cell (WBC) ≥ 3.5×10*9/L; neutrophil count (NEUT) ≥ 1.5×10*9/L; platelets (PLT) ≥ 100×10*9/L; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5×UNL; total bilirubin (TBIL) ≤ 1.5×UNL; creatinine ≤ 1.5UNL; blood urea nitrogen (BUN) ≤ 1.0×UNL.

Exclusion Criteria:

1. Synchronous and metachronous primary malignancies in but not limited to the upper aerodigestive tract, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix.
2. Patients have undergone any type of anti-cancer treatment.
3. Baseline clinical stage M1 per AJCC 8th edition of staging classification, including supraclavicular lymph node metastases.
4. Investigators assessed major vessel involvement with high-risk hemorrhage.
5. A higher probability of esophageal perforation during conversion therapy.
6. Active infectious diseases, including but not limited to tuberculosis, hepatitis B virus, or hepatitis C virus.
7. Allergic to anti-cancer agents, including but not limited to anti-PD-1 or chemotherapy agents.
8. Given cardiopulmonary dysfunction, patients can not tolerate conversion therapy or surgery.
9. Pregnant or lactating women and women of childbearing potential who lacked effective contraception.
10. Non-compliance with the inclusion criteria judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 4 months
  Minimal distance tumor/circumferential resection margin (CRM) > 1 mm.

SECONDARY OUTCOMES:
1-year OS rate | 1 year after all treatment
  Defined as the proportion of patients still alive within one year from treatment initiation.
1-year PFS | 1 year after all treatment
  Defined as the proportion of patients without disease progression or death within one year from treatment initiation.
Positive rate of circulating tumor DNA (ctDNA) in minimal residual disease (MRD) before and after neoadjuvant treatment and its correlation with the pathological response and disease progression during surveilance | 6 month
  To investigate whether ctDNA variation can be used for MRD predicting incidence of pathological incidence and monitoring tumor progression after surgery
Incidence of Treatment-Emergent Adverse Events | 4 month
  Adverse event during chemoRT or immunotherapy
Pathological response rate | 4 month
Postoperative complications | 4 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, National Cancer Center, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China

IPD SHARING:
Plan to Share IPD: No